CLINICAL TRIAL: NCT04057027
Title: The Effect of Delayed Cord Clamping and Milking on the Amount of Endogenous Stem Cells In Preterm Infants
Brief Title: The Effect of Delayed Cord Clamping and Milking on the Amount of Stem Cells In Preterm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Collaborators: Turkish Neonatology Society (Other)
Responsible Party: Principal Investigator, Merih Cetinkaya, Neonatologist, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: KAEK/2019.02.36
Record Dates: First submitted 2019-05-15; First posted 2019-08-14 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Umbilical Cord; Clamping Time
MeSH Terms: interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Delayed Cord Clamping for 30 seconds (Experimental): Infants whose umbilical cord clamping will be delayed for 30 secs.
  Interventions: Procedure: Delayed umbilical cord clamping
- Delayed Cord Clamping for 60 seconds (Experimental): Infants whose umbilical cord clamping will be delayed for 60 secs.
  Interventions: Procedure: Delayed umbilical cord clamping
- Umbilical Cord Milking (Experimental): Infants whose umbilical cord will be clamped after milking from the distance of 20 cm from mother's side to the baby for 3-4 times.
  Interventions: Procedure: Cord Milking

INTERVENTIONS:
Procedure: Delayed umbilical cord clamping — During the C section, infants' umbilical cord clamping will be delayed for 30-60 seconds.
  Arms: Delayed Cord Clamping for 30 seconds; Delayed Cord Clamping for 60 seconds
Procedure: Cord Milking — Umbilical cord will be milked from th distance of 20cm from mother's side to the baby, for 3-4 times.
  Arms: Umbilical Cord Milking

SUMMARY:
Stem cell therapies have been promising therapies in neonatal morbidities such as bronchopulmonary dysplasia, intraventricular hemorrhage and hypoxic ischemic encephalopathy. Although researchers showed those effects by several mechanisms including paracrine effect, regenerative and restorative effects, there is no obvious recommendations for the type of stem cells, dosage or the route of administration the cells. The usage of exogenous stem cells can be difficult due to technical issues in preterm infants.

In the presence of these data, the amount of endogenous stem cells passing through the cord to the infant may show differences in terms of delayed cord clamping and milking. Therefore the aim of this prospective randomized study is to determine the quantity of the stem cells according to delayed cord clamping or cord milking. We also aimed to evaluate the association between the number of stem cells and neonatal morbidities.

ELIGIBILITY:
Inclusion Criteria:

* Infants born under 32 weeks of gestation
* Accepted to participate with informed consent
* History of healthy pregnancy
* Infants born and will be followed up at the study hospital

Exclusion Criteria:

* Congenital abnormalities
* Chromosomal abnormalities
* Declined to participate

Max Age: 30 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-09-05 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of Stem cells | 6 months
  Determining the quantity of endogenous stem cells transmitted through the umbilical cord to the infant after different types of cord clamping.

SECONDARY OUTCOMES:
Number of Participants with Neonatal Morbidities | 6 months
  Recording newborn morbidities such as intraventricular hemorrhage , necrotizing enterocolitis, bronchopulmonary dysplasia , retinopathy of prematurity which are detected in the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Yilmaz Semerci, Principal Investigator — Kanuni Sultan Süleyman Eah
Locations (1):
- Istanbul Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No